CLINICAL TRIAL: NCT04597697
Title: A Trial Investigating the Pharmacokinetic Properties of Insulin Icodec in Subjects With Various Degrees of Hepatic Impairment
Brief Title: A Study to Test How a New Long-acting Insulin (Insulin Icodec) Works in the Body of People With Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4570
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects with normal hepatic function (Experimental): The participants will be allocated into four groups. Receiving one insulin icodec dose, administered subcutaneously.
  Interventions: Drug: Insulin icodec
- Subjects with mild hepatic impairment, child-pugh grade A (Experimental): The participants will be allocated into four groups. Receiving one insulin icodec dose, administered subcutaneously.
  Interventions: Drug: Insulin icodec
- Subjects with moderate hepatic impairment, child-pugh grade B (Experimental): The participants will be allocated into four groups. Receiving one insulin icodec dose, administered subcutaneously.
  Interventions: Drug: Insulin icodec
- Subjects with severe hepatic impairment, child-pugh grade C (Experimental): The participants will be allocated into four groups. Receiving one insulin icodec dose, administered subcutaneously.
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: Insulin icodec — Insulin icodec will be investigated in participants with impaired liver function and subjects with normal liver function. Administered as a single dose subcutaneously (under the skin) The study will last for about 8 weeks.

SUMMARY:
Participants will receive one insulin icodec dose, which will be administered in the morning of the day of dosing.

The study will last for about 8 weeks. Participants will have 8 visits with the study doctor in the clinical research unit.

Insulin icodec will be injected into a skin fold with a small needle (subcutaneous application) using a pen injector prefilled with a volume of 3 mL (about a spoonful).

Participants must not participate if they meet certain conditions called exclusion criteria, such as an age of below 18 years or above 70 years, if participants are over- or underweight, using certain medicines, or have serious health conditions (other than impaired liver function ).

Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-70 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.5 and 39.9 kg/m^2 (both inclusive) Specific inclusion criterion only for subjects with hepatic impairment
* Subjects with stable hepatic impairment classified as Child-Pugh grade A, B or C as assessed by the investigator. Stable hepatic impairment is defined as no clinically significant change in disease status, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)
* Diagnosis of diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
AUC,Ico,0-inf,SD, Area under the serum insulin icodec concentration-time curve after a single dose | Day 1
  From 0 hours until infinity after trial product administration (pmol*h/L)

SECONDARY OUTCOMES:
Cmax,Ico,SD, Maximum observed serum insulin icodec concentration after a single dose | Day 1
  From 0 hours until last measurement time after trial product administration (pmol/L)
tmax,Ico,SD, Time to maximum observed serum insulin icodec concentration after a single dose | Day 1
  From 0 hours until last measurement time after trial product administration (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Czechia
- Summit Clinical Research s.r.o., Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Haahr H, Cieslarova B, Hingst JR, Jiang S, Kristensen NR, Kupcova V, Norgreen L, Wagner FH, Ignatenko S. The Effect of Various Degrees of Renal or Hepatic Impairment on the Pharmacokinetic Properties of Once-Weekly Insulin Icodec. Clin Pharmacokinet. 2024 Jun;63(6):819-830. doi: 10.1007/s40262-024-01375-2. Epub 2024 May 9. PMID 38722461